CLINICAL TRIAL: NCT00025571
Title: A Phase I Study of Photodynamic Therapy (PDT) Using 2-(1-hexyloxyethyl)-2 Devinyl Pyropheophorbide-a (HPPH) for Treatment of Early Stage Lung Cancer - A Dose Ranging Study
Brief Title: Photodynamic Therapy With HPPH in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Gregory Loewen, MD, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000068974; RPCI-RP-0005
Record Dates: First submitted 2001-10-11; First posted 2003-06-25 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: HPPH

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make tumor cells more sensitive to light to kill tumor cells. Photosensitizing drugs such as HPPH are absorbed by tumor cells and, when exposed to light, become active and kill the tumor cells.

PURPOSE: Phase I trial to study the effectiveness of photodynamic therapy with HPPH in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the systemic and normal tissue toxicity of photodynamic therapy with HPPH in patients with early stage or centrally obstructing non-small cell lung cancer.
* Determine, preliminarily, the efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of HPPH.

Patients receive HPPH IV over 1 hour on day 1. Patients undergo laser light therapy via bronchoscopy on day 3.

Cohorts of 3-6 patients receive escalating doses of HPPH until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for at least 6 months.

PROJECTED ACCRUAL: Approximately 15-17 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed microinvasive or centrally obstructing non-small cell lung cancer

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Large cell carcinoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100% OR
* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL
* Alkaline phosphatase no greater than 3 times upper limit of normal (ULN)
* SGOT no greater than 3 times ULN
* PT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 3.0 mg/dL

Pulmonary:

* No severe chronic obstructive pulmonary disease that would preclude study

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No contraindications to bronchoscopy
* No porphyria
* No hypersensitivity to porphyrin or porphyrin-like compounds

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy for lung cancer allowed

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Prior endocrine therapy for lung cancer allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent external beam radiotherapy

Surgery:

* No concurrent surgery

Other:

* Prior therapy for lung cancer allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2002-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M. Loewen, DO, FCCP, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States